CLINICAL TRIAL: NCT02486926
Title: The Effects of Remifentanil and Remifentanil-Alfentanil Administration on Emergence Agitation After Brief Ophthalmic Surgery in Children
Brief Title: The Effects of Remifentanil and Remifentanil-Alfentanil Administration in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-I069
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Adverse Effect of Other General Anesthetics
MeSH Terms: interventions — Sevoflurane; Remifentanil; Alfentanil; Thiopental; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Sevoflurane (Placebo Comparator): Anesthesia was maintained with sevoflurane,and the incidence and severity of emergence agitation was investigated.
  Interventions: Other: Sevoflurane; Drug: Thiopental; Drug: Rocuronium
- Remifentanil (Active Comparator): Anesthesia was maintained with sevoflurane and remifentanil. The incidence and severity of emergence agitation was compared with sevoflurane group.
  Interventions: Other: Sevoflurane; Drug: Remifentanil; Drug: Thiopental; Drug: Rocuronium
- Alfentanil (Active Comparator): Anesthesia was maintained with sevoflurane and remifentanil, and alfentanil was administered 10 min before the end of surgery.
  The incidence and severity of emergence agitation was compared with sevoflurane group.
  Interventions: Other: Sevoflurane; Drug: Remifentanil; Drug: Alfentanil; Drug: Thiopental; Drug: Rocuronium
- Thiopental (Other): General anesthesia was induced with thiopental 5 mg/kg, rocuronium 0.6 mg/kg and sevoflurane in all patients.
  Interventions: Other: Sevoflurane; Drug: Remifentanil; Drug: Alfentanil; Drug: Thiopental; Drug: Rocuronium
- Rocuronium (Other): General anesthesia was induced with thiopental 5 mg/kg, rocuronium 0.6 mg/kg and sevoflurane in all patients.
  Interventions: Other: Sevoflurane; Drug: Remifentanil; Drug: Alfentanil; Drug: Thiopental; Drug: Rocuronium

INTERVENTIONS:
Other: Sevoflurane — Anesthesia of patients was maintained only with sevoflurane.
Drug: Remifentanil — Anesthesia of patients was maintained with both sevoflurane and continuous remifentanil infusion.
  Other Names: Ultiva
  Arms: Alfentanil; Remifentanil; Rocuronium; Thiopental
Drug: Alfentanil — Anesthesia was maintained with both sevoflurane and continuous infusion of remifentanil. Alfentanil was administrated (5ug/kg) to patients 10 minutes before the end of surgery.
  Arms: Alfentanil; Rocuronium; Thiopental
Drug: Thiopental — General anesthesia was induced with thiopental 5 mg/kg, rocuronium 0.6 mg/kg and sevoflurane in all patients.
  Other Names: Pentothal sodium
Drug: Rocuronium — General anesthesia was induced with thiopental 5 mg/kg, rocuronium 0.6 mg/kg and sevoflurane in all patients.
  Other Names: Esmeron

SUMMARY:
Sevoflurane is widely and frequently used in pediatric anesthesia due to its non-irritating airway properties, rapid induction and emergence. However, it is associated with emergence agitation (EA) in children. EA may cause injury to the child or to the surgical site and is a cause of stress to both caregivers and families. Various pharmacologic agents have been suggested to reduce EA. But the effect of remifentanil on EA is still controversial. This study was designed to compare the effects of remifentanil and remifentanil combining alfentanil on EA in children undergoing ophthalmic surgery with sevoflurane anesthesia.

DETAILED DESCRIPTION:
One hundred and two children, aged 3-9 years, undergoing ophthalmic surgery were studied. General anesthesia was induced with thiopental 5 mg/kg, rocuronium 0.6 mg/kg and sevoflurane. At the time of separation from parents, separation score was recorded. When the children have a separation score of three or four point, they received half dose of thiopental before going to the operation room. They randomly assigned to group S (sevoflurane alone) or group R (sevoflurane with remifentanil infusion at the rate of 0.1 ㎍/kg/min) or group A (sevoflurane with remifentanil infusion and intravenous injection of alfentanil 5 ㎍/kg 10 min before the end of surgery). Mean arterial pressure (MAP), heart rate (HR) and sevoflurane concentration were checked every 15 minutes after induction of anesthesia. Time to extubation from discontinuation of sevoflurane inhalation was measured. Time to discharge from postanesthesia care unit (PACU) was assessed with postanesthetic Aldrete recovery score. Emergence agitation scoring system was used to evaluate the incidence and severity of EA.

ELIGIBILITY:
Inclusion Criteria:

* children who were scheduled to undergo ophthalmic surgery under general anesthesia

Exclusion Criteria:

* developmental delay, neurologic or psychologic disease,
* history of sleep apnea,
* or history of general anesthesia

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
the incidence of emergence agitation | during recovery time in PACU (within 1 hour)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kyung Lee, M.D., Study Chair — Department of Anesthesiology and Pain Medicine, Hallyum University Sacred Heart Hospital

REFERENCES:
- [Background] Ozturk T, Erbuyun K, Keles GT, Ozer M, Yuksel H, Tok D. The effect of remifentanil on the emergence characteristics of children undergoing FBO for bronchoalveolar lavage with sevoflurane anaesthesia. Eur J Anaesthesiol. 2009 Apr;26(4):338-42. doi: 10.1097/EJA.0b013e32831de50d. PMID 19401665
- [Derived] Choi YH, Kim KM, Lee SK, Kim YS, Kim SJ, Hwang WS, Chung JH. Effects of remifentanil and remifentanil-alfentanil administration on emergence agitation after brief ophthalmic surgery in children. BMC Anesthesiol. 2016 Aug 2;16(1):50. doi: 10.1186/s12871-016-0213-2. PMID 27484339